CLINICAL TRIAL: NCT05931484
Title: A Phase 2, Double-Blind, Multi-Center, Placebo-Controlled Clinical Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of FHL-301 in Adult Patients With Parkinson's Disease
Brief Title: Study to Evaluate the Safety, Tolerability, Efficacy, and PK of FHL-301 in Parkinson's Disease Patients.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Hills Lab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHL-301-001
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Gemfibrozil

STUDY DESIGN:
Intervention Model Description: This is a phase 2, double-blind, multi-center, placebo-controlled clinical study to evaluate the safety, tolerability, efficacy, and PK of FHL-301 in adult patients with early-stage PD. Following screening, qualifying patients who meet all inclusion and exclusion criteria will be randomized 1:1 ratio to receive FHL-301 or Placebo. The study is comprised of two phases: the Dose Titration Phase (DTP) in which participants will be started with a dose of 200 mg BID (30 minutes before the morning and evening meals) and increased during a 3-week treatment period. Patients who complete the DTP of the study will enter the Maintenance Phase and remain on the final titrated dose for up to 48 weeks post titration. If at any stage during the titration phase the participant cannot tolerate the increased dose, the dose will be decreased by 100 mg BID weekly until the highest tolerated dose is reached.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Active
  Interventions: Drug: Gemfibrozil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemfibrozil — Oral Solution
  Arms: Active
Drug: Placebo — Daily dose of Placebo
  Other Names: Placebo to match Gemfibrozil solution
  Arms: Placebo

SUMMARY:
This is a phase 2, double-blind, multi-center, placebo-controlled clinical study to evaluate the safety, tolerability, efficacy, and PK of FHL-301 in adult patients with early-stage PD. Following screening, qualifying patients who meet all inclusion and exclusion criteria will enter the study and be randomized 1:1 to receive FHL-301 or Placebo at a starting dose of 200 mg BID (30 minutes before the morning and evening meals) during the 3-week titration period. To determine the tolerance of each participant for FHL-301, titration will increase by 200 mg BID every week until the maximum dose of 600 mg BID or the highest tolerated dose of 1200 mg daily is reached and maintained for 1 week. Thereafter, patients who complete the dose Titration Phase of the study will enter the Maintenance Phase and remain on the final titrated dose for up to 48 weeks post titration. If at any stage during the titration phase the participant cannot tolerate the increased dose, the dose will be decreased by 100 mg BID weekly until the highest tolerated dose is reached.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must fulfill the following inclusion criteria:

  * A diagnosis of clinically established PD in accordance with the Movement Disorder Society (MDS) ClinicalDiagnostic Criteria for PD (Confirmed by DaTscan).
  * Each patient must be able and willing to provide signed and dated informed consent prior to the study.
  * Female and male patients 40 to 75 years of age inclusive.
  * Female patients of childbearing potential must not be pregnant or lactating with a negative serum human chorionic gonadotropin (HCG) pregnancy test result at Screening.
  * Female patients of childbearing potential and male patients must use an adequate method of contraception from Screening until completion of the study. Acceptable methods of contraception are barrier methods (male condom, female condom, diaphragm, cervical cap, spermicide, or intrauterine device [IUD]), surgical sterility (documented doctor's report of vasectomy, hysterectomy, and/or bilateral oophorectomy), and/or postmenopausal status (defined as at least 1 year without menses as demonstrated by medical history or patient report).
  * Treatment naïve patients for PD
  * Hoehn and Yahr Stage of 1.0 to 2.0 at Screening

Exclusion Criteria:

* Diagnosis is unclear, or a suspicion of other Parkinsonian syndrome exists, such as secondary Parkinsonism (caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), Parkinson-plus syndromes, or Huntington's disease.
* The presence of a clear diagnosis of neurodegenerative diseases other than PD
* Have undergone surgery for the treatment of PD (e.g., pallidotomy, deep brain stimulation, fetal tissue transplantation) or have undergone any other brain surgery at any time, even for non-PD conditions.
* Current/history of psychiatric diagnosis of acute psychotic disorder or other primary psychiatric diagnoses, i.e., bipolar disorder or MDD, or other psychiatric, neurological or behavioral disorders/symptoms that may interfere with conduct of study.
* Montreal Cognitive Assessment (MoCA) score < 23
* Clinical chemistry assessments that indicate clinically significant major or unstable disease such as: abnormal white or red blood cell count; aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) above 3x the upper limit of normal; or estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
* Pre-existing diagnosis of gastrointestinal diseases which may hamper absorption of study medication, such as liver and gallbladder diseases (e.g., cholangitis and cholestasis), Crohn's disease or ulcerative colitis.
* Female participants that are pregnant or planning to become pregnant.
* Significant neurologic disease such as AD, stroke, brain tumor, multiple sclerosis or seizure disorder.
* Major depression in past 12 months (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-5] criteria), major mental illness such as schizophrenia, or recent (in past 12 months) alcohol or substance abuse.
* Use of any investigational agents within 30 days prior to screening.
* Sensitivity, intolerance, or allergies to FHL-301.
* Patient with any history or current evidence of suicidal ideation in the last year.
* Unwilling to complete any planned study assessments.
* Any contraindication for undergoing a Magnetic resonance imaging (MRI) scan of the head.
* Abnormal MRI findings in the mega cisterna, septum pellucidum, signs of severe cortical or subcortical atrophy, brain tumors, vascular diseases, trauma or arteriovenous malformations
* Patient has any additional illnesses that in the Investigator's opinion would cause them to be at risk with treatment with FHL-301.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2027-11-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale | 52 weeks
  Change from Baseline in the Unified Parkinson's Disease Rating Scale Part III (motor examination) at maintenance Week 48 in the modified Full Analysis Set (mFAS) population.
  * Motor : range 0-132
  * 32 and below is mild and 59 and above is severe.